CLINICAL TRIAL: NCT02567006
Title: SMS Mobile Technology to Improve Early Childhood Vaccine Coverage in Guatemala
Acronym: SMSVaxGuate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Universidad del Valle, Guatemala (Other); Fundacion para la Salud Integral de los Guatemaltecos CU (Other); Ministry of Health, Guatemala (Other Government); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 14-2170; 1R21HD084115-01 (NIH)
Record Dates: First submitted 2015-09-30; First posted 2015-10-02 (Estimated); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Adherence to Vaccination Schedules; Timeliness of Vaccination; Acceptability of SMS Reminder Program
Keywords: vaccines; reminders; immunization timeliness; vaccine coverage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Short Message Service (SMS) group (Active Comparator): Receiving SMS message reminders 1 week before scheduled vaccination
  Interventions: Behavioral: SMS message
- Usual care (Placebo Comparator): Not receiving SMS messages
  Interventions: Other: Usual care

INTERVENTIONS:
Behavioral: SMS message — SMS messages will be delivered at 6, 4, and 2 days before the next scheduled date of the primary vaccines for the intervention group
  Other Names: text messages
  Arms: Short Message Service (SMS) group
Other: Usual care — Health clinic nurse provides regular appointment in the vaccination card with no active reminders
  Arms: Usual care

SUMMARY:
This project plans to learn more about whether sending text messages to parents on their mobile phones to remind them when their child is due for his or her next vaccination will improve children getting vaccinated on time.

DETAILED DESCRIPTION:
This project plans to learn more about whether sending text messages to parents on their mobile phones to remind them when their child is due for his or her next vaccination will improve children getting vaccinated on time. The vaccines that will be given are the same routine vaccinations registered in Guatemala and used by the Ministry of Health regardless of enrollment in the study.

ELIGIBILITY:
Inclusion Criteria:

* First dose of primary vaccination series
* Parents owning a mobile phone and able to decipher SMS messages
* Consent form signed

Exclusion Criteria:

* Moving away from the study site in the next 12 months
* Ineligible for primary vaccination series by the MOH

Ages: 6 Weeks to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 720 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2017-07-07 (Actual); Study Completion 2017-07-10 (Actual)

PRIMARY OUTCOMES:
Completion of vaccine primary series | 12 months of age
  Completion of 2nd and 3rd dose of vaccines by 1 year of age

SECONDARY OUTCOMES:
Factors associated with immunization delays | 12 months
  Demographic, education and behavioral factors associated with days late for vaccination
Acceptability of SMS vaccine reminders | 12 months
  Qualitative data from focus groups to evaluate acceptability of SMS program
Timeliness of immunization | 12 months
  Days delayed from date for 2nd and 3rd dose of vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Edwin J Asturias, MD, Study Chair — University of Colorado, Denver; Gretchen Domek, MD, Principal Investigator — University of Colorado, Denver; Ingrid L Contreras, MD, Study Director — University del Valle, Guatemala
Locations (2):
- Guatemala (2):
  - Fundacion para la Salud Integral de los Guatemaltecos CU, Coatepeque, Departamento de Quetzaltenango
  - University del Valle, Guatemala, Guatemala City

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gurman TA, Rubin SE, Roess AA. Effectiveness of mHealth behavior change communication interventions in developing countries: a systematic review of the literature. J Health Commun. 2012;17 Suppl 1:82-104. doi: 10.1080/10810730.2011.649160. PMID 22548603
- [Background] Head KJ, Noar SM, Iannarino NT, Grant Harrington N. Efficacy of text messaging-based interventions for health promotion: a meta-analysis. Soc Sci Med. 2013 Nov;97:41-8. doi: 10.1016/j.socscimed.2013.08.003. Epub 2013 Aug 13. PMID 24161087
- [Derived] Palmer MJ, Henschke N, Bergman H, Villanueva G, Maayan N, Tamrat T, Mehl GL, Glenton C, Lewin S, Fonhus MS, Free C. Targeted client communication via mobile devices for improving maternal, neonatal, and child health. Cochrane Database Syst Rev. 2020 Jul 14;8(8):CD013679. doi: 10.1002/14651858.CD013679. PMID 32813276
- [Derived] Domek GJ, Contreras-Roldan IL, Bull S, O'Leary ST, Bolanos Ventura GA, Bronsert M, Kempe A, Asturias EJ. Text message reminders to improve infant immunization in Guatemala: A randomized clinical trial. Vaccine. 2019 Sep 30;37(42):6192-6200. doi: 10.1016/j.vaccine.2019.08.046. Epub 2019 Sep 3. PMID 31492475
- [Derived] Domek GJ, O'Leary ST, Bull S, Bronsert M, Contreras-Roldan IL, Bolanos Ventura GA, Kempe A, Asturias EJ. Measuring vaccine hesitancy: Field testing the WHO SAGE Working Group on Vaccine Hesitancy survey tool in Guatemala. Vaccine. 2018 Aug 23;36(35):5273-5281. doi: 10.1016/j.vaccine.2018.07.046. Epub 2018 Jul 27. PMID 30061026